CLINICAL TRIAL: NCT02481570
Title: Evaluation of an Anesthetic Optimization Technique in Adolescent Idiopathic Scoliosis Surgery
Brief Title: Anesthetic Optimization in Scoliosis Surgery
Acronym: AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201500120
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Adolescent Idiopathic Scoliosis; Respiratory Depression; Postoperative Pain
Keywords: Adolescent Idiopathic Scoliosis; Scoliosis surgery; Pharmacokinetic simulation
MeSH Terms: conditions — Respiratory Insufficiency; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anesthesia optimization (Experimental): Information from the pharmacokinetic simulation during an anesthetic regimen of a propofol based Total Intravenous Anesthetic (TIVA)
  Interventions: Other: pharmacokinetic simulation

INTERVENTIONS:
Other: pharmacokinetic simulation — The aim of the simulation is to recommend dosing adjustments to improve postoperative analgesia with a rapid emergence.

SUMMARY:
The standard anesthetic care plan for people having adolescent idiopathic scoliosis surgery will be accompanied by a pharmacokinetic simulation of the administered drugs to suggest opportunities to adjust drug doses to achieve tolerable pain control after surgery, avoid respiratory depression and allow patients to respond quickly either during intraoperative testing or at the conclusion of surgery.

DETAILED DESCRIPTION:
As part of this study, anesthesiologists will be given additional data on the expected drug effects based on a computer simulation. The data will be provided as a suggestion and will be used together with all the other information normally used to keep the study subjects safely asleep during surgery. In addition, data will be collected from the medical history and on postoperative pain control and medication side effects for the first 24 hours. Specifically, study subjects will be asked to rate their pain on a 10-point scale after they wake up from surgery and once they arrive in the pediatric intensive care unit. Measures of the time from the end of surgery until the study subjects are awake and out of the operating room will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 1-2
* At least 10 years of age and not older than 18 years of age
* Diagnosis of idiopathic adolescent scoliosis

Exclusion Criteria:

* Currently pregnant
* Currently breastfeeding
* Currently being treated with opiates
* Currently being treated with alpha2 agonists
* Currently being treated with anticonvulsants
* Currently being treated with antidepressants
* History of significant restrictive lung disease

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
4-Item Pain Intensity Measure | 24 hours
  0 - 10 (0=no pain; 10 = pain as bad as can be)
Respiratory depression | 24 hours
  Respiratory rate less than 10 breaths per minute (bpm), or administration of naloxone.

SECONDARY OUTCOMES:
Utility of pharmacokinetic simulation | 4 - 8 hours (Intraoperative period)
  The number of modifications to the anesthetic dosing

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Seubert, MD PhD DABNM, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tams C, Dooley FC, Sangari TS, Gonzalez-Rodriguez SN, Stoker RE, Phillips SA, Koenig M, Wishin JM, Molinari SC, Blakemore LC, Seubert CN. Methadone and a Clinical Pathway in Adolescent Idiopathic Scoliosis Surgery: A Historically Controlled Study. Global Spine J. 2020 Oct;10(7):837-843. doi: 10.1177/2192568219878135. Epub 2019 Sep 26. PMID 32905725